CLINICAL TRIAL: NCT01089608
Title: Efficacy and Safety Assessment of Azyter® Eye Drops (T1225) in Patients With Blepharitis (Pilot Phase II Clinical Study, Multicentre, Randomised, Double Masked, Comparative, 2 X 40 Patients)
Brief Title: Efficacy and Safety Assessment of Azyter® Eye Drops (T1225) in Patients With Blepharitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Collaborators: Keyrus Biopharma (Other); VEEDA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LT1225-PII-06/09; 2009-017388-41 (EudraCT Number)
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Blepharitis
Keywords: Azyter in patients affected by chronic blepharitis.
MeSH Terms: conditions — Blepharitis | interventions — Azithromycin; Povidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unifluid (Placebo Comparator): Eye drops in Single Dose Unit
  Interventions: Drug: Povidone
- Azithromycin (Experimental): Eye drops Single dose unit
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Eye drops, Dosage : 1.5%
  1 drop twice daily at Day 0, then 1 drop once daily from Day 1 to Day 6 in the morning, following by a period of 2 weeks without treatment. This therapeutic scheme will be repeat 2 times.
  Other Names: T1225 1.5% - Azyter -
  Arms: Azithromycin
Drug: Povidone — Eye drops Single dose unit
  1 drop twice daily at Day 0, then 1 drop once daily from Day 1 to Day 6 in the morning, following by a period of 2 weeks without treatment. This therapeutic scheme will be repeat 2 times.
  Other Names: Unifluid
  Arms: Unifluid

SUMMARY:
The primary objective of this study is to demonstrate the efficacy of T1225 eye drops versus placebo eye drops on the global ocular discomfort (VAS).

DETAILED DESCRIPTION:
Currently, topical antibiotic ointments are used for blepharitis. They provide prolonged contact time with the lid margin but with little penetration into eyelid tissue. Azithromycin eye drops may offer on advantage over these preparations because azithromycin achieves sustained high concentration in various ocular tissues including the lid margin.

Patients will be treated during 7 days (1 drop twice daily the first day following by one drop once daily for 6 days) following by a period of 2 weeks without treatment. This therapeutic scheme will be repeated two times.

Efficacy will be evaluated by change from baseline (Day 0) to Day 63 Â± 3 Days of the global ocular discomfort evaluation (VAS).

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of moderate to severe chronic blepharitis (posterior and/or anterior) in at least one eligible eye

Exclusion Criteria:

* Monophtalmia
* Eyelid dysfunction
* Facial paralysis.
* Severe dry eye syndrome.
* Ocular metaplasia.
* Filamentous keratitis
* Schirmer test < 5 mm.
* Best far corrected visual acuity < 1/10.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe BAUDOUIN, Professor, Principal Investigator
Locations (1):
- C.H.N.O des XV-XX, Paris, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Unifluid: Eye drops in Single Dose Unit
  Povidone: Eye drops Single dose unit
  1 drop twice daily at Day 0, then 1 drop once daily from Day 1 to Day 6 in the morning, following by a period of 2 weeks without treatment. This therapeutic scheme will be repeat 2 times.
- Azithromycin: Eye drops Single dose unit
  Azithromycin: Eye drops, Dosage : 1.5%
  1 drop twice daily at Day 0, then 1 drop once daily from Day 1 to Day 6 in the morning, following by a period of 2 weeks without treatment. This therapeutic scheme will be repeat 2 times.
Period: Overall Study
Arm/Group | Unifluid | Azithromycin
Started | 43 | 50
Completed | 43 | 44
Not Completed | 0 | 6
Not completed — Adverse Event | 0 | 4
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unifluid | Azithromycin | Total
Number analyzed (Participants) | 43 | 50 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (16.2) | 55.7 (16.1) | 56.2 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 17 | 25 | 42

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS - Ranges 0-100 mm)
Description: The primary objective is to evaluate the efficacy of the treatment by the change from baseline (Day 0) to Day 63 (± 3 Days) of the global ocular discomfort (Visual Analogue Scale) (Decrease of VAS value = better outcome)
Time Frame: Baseline and D63 (D63 minus baseline)
Population: Modified ITT set: all randomised patients with at least one eligible treated eye, for whom any follow-up efficacy data are available.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale (from 0 to 100 mm)
Arm/Group | Unifluid | Azithromycin
Number analyzed (Participants) | 43 | 50
units on a scale (from 0 to 100 mm) | 36.5 [30.5 to 42.4] | 28.5 [22.7 to 34.3]
Statistical Analysis 1: Comparison: Unifluid vs Azithromycin; Test type: Superiority or Other; p = 0.072, Mixed Models Analysis; Mean Difference (Net) = -8.01, 95% CI 2-sided [-16.30 to 0.28]

ADVERSE EVENTS:
Arm/Group | Unifluid | Azithromycin
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/50
Other Adverse Events (participants affected / at risk) | 0/43 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the results of the Trial are the sole and exclusive property of THEA, and cannot be used in whatever form without prior written agreement of THEA.